CLINICAL TRIAL: NCT02037685
Title: Improving Adherence to Cholesterol Lowering Medications Among Minority Populations in Florida: A Randomized Trial
Brief Title: Improving Adherence to Statins Among Minority Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Humana Inc. (Industry)
Responsible Party: Principal Investigator, Ana M. Palacio, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1KG11; 4KB13 (Other Grant/Funding Number: James and Esther King BIomedical Research Program)
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Dyslipidemia
Keywords: Statins; Cholesterol lowering medications; Adherence; Motivational interviewing; Minority populations
MeSH Terms: conditions — Dyslipidemias | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Subjects randomized to usual care will receive a brochure once a year on the importance and impact of controlling cardiovascular risk factors, tips to improve statin adherence and smoking cessation strategies and public services. Subjects will also receive a letter every 6 months to remind about study participation along with educational material.
  Interventions: Other: Usual Care
- Motivational Interviewing (MINT) (Experimental): The MINT intervention will consist of 6 to 9 telephone encounters between a counselor trained in Motivational interviewing. All subjects in the MINT arm will be contacted every 3 months; however subjects who are not filling medication appropriately will receive additional calls.
  Each telephone encounter will last from 20 to 30 minutes and have a patient centered approach having the following basic structure and goals:
  * Establishing a connection and reinforcing autonomy: .
  * Empathizing with ambivalence and rolling with resistance.
  * Coach the subject towards expressions of commitment.
  Interventions: Behavioral: Motivational Interviewing (MINT)

INTERVENTIONS:
Behavioral: Motivational Interviewing (MINT) — MINT has the following basic structure and goals:
  * Establishing a connection and reinforcing autonomy: open ended questions regarding the health status or well being of the participant to establish an empathetic connection with the subject via reflective listening.
  * Empathizing with ambivalence and rolling with resistance. The counselor will help the subject express the ambivalence they may have regarding taking their statins.
  * Coach the subject towards expressions of commitment. Commitment is predictive of change. Speaking commitment out loud to an "other" enhances the likelihood that the commitment will be acted upon
  Arms: Motivational Interviewing (MINT)
Other: Usual Care — We selected American Heart Association brochures on a variety of risk factors, including dyslipidemia and mailed them to subjects in the usual care.
  Arms: Usual care

SUMMARY:
Statins are cholesterol lowering medications that reduce the risk of cardiovascular events. However adherence to these medications has been found to be lower among minorities, a group particularly vulnerable for heart disease.

The purpose of this study is to compare the efficacy of a phone based behavioral intervention to mailed educational materials regarding how to control cholesterol and other risk factors. We hypothesized that the behavioral intervention will improve adherence to statins by 15%.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) disproportionately affects members of certain racial/ethnic minority groups.Further in spite of a reduction in rates of cardiovascular events,the gap between certain minority groups and non-minority groups has not diminished. Cholesterol lowering medications are a medically proven intervention that dramatically reduces the risk of primary and secondary cardiovascular outcomes.However, the literature shows that at one year only half of the patients prescribed this medication continue to take a statin. One well known risk factor shown to be a predictor for non adherence is belonging to a racial/ ethnic minority group.

The focus of the proposed study is to examine a non-traditional care-management approach delivered by a large commercial health benefit carrier in the prevention of cardiovascular disease among minority populations who have cardiovascular risk factors and who have been started in cholesterol lowering therapy. In particular, we seek to determine if a culturally tailored phone based intervention (Motivational Interviewing) delivered to Latino and African American enrollees living in predominantly minority neighborhoods in Florida, is effective at improving adherence to Statins.

Specific Aims

1. To prospectively identify 1200 Latino or African American residing in Florida who have received a new prescription for statin therapy, evaluate their adherence to the statin and determine if the reasons for non-adherence are similar or different from other studies of adherence to cardiovascular medications.
2. Conduct a randomized control trial to compare the effectiveness of a motivational interviewing telephonic intervention to usual care on the primary outcome of statin adherence among minority subjects living in Florida.

In addition, among the tobacco users at baseline we will evaluate the impact of our phone based MINT intervention on tobacco cessation in this minority populations.

Update: The sponsor and the IRB approved a reduction in the target number of participants to 800. The reason was that we experienced a recruitment delay to ensure HIPAA compliant procedures between the University and the Health Benefits company when the Humana research group moved out of the University campus. Data that became available from another study showed 800 subjects will yield enough power for the analyses planned originally.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over age 35 years
2. Recent new prescription for a Statin (GPI code 39.40.xx ) which will be the index prescription. We will define new as no GPI code present for any statin over a 6 month period before the index prescription.
3. Self report of being Latino or AA.

Exclusion Criteria:

* Enrollment in any other CVD intervention program

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 779 (Actual)
Dates: Start 2010-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Medication possession ratio (MPR) | 12 months after the statin prescription
  The primary outcome will be MPR for statin medication equal or above .80. MPR is a continuous multiple interval measure of medication availability. The medication possession ratio is defined as the sum of the days' supply of medication divided by the number of days between the enrollment and the last day of follow up. The binary dependent variable is: MPR equal to or above .80 (adequate adherence or drug availability during 80% or more of the therapy time) and MPR below .80 (non adherence or drug availability during less than 80% of the therapy time).

SECONDARY OUTCOMES:
Self-reported adherence score (Morisky Medication Adherence Scale-8) | At baseline and 12 months after statin prescription
  8-item questionaire to measure self reported adherence to statin

OTHER OUTCOMES:
Smoking status | At baseline and at 12 months
  Smoking history questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Ana Palacio, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The IRB application did not include the use of the data for future research